CLINICAL TRIAL: NCT07135843
Title: iPATH - Digital Home-Based Training for Physical Activity Promotion in Older Adults After Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Digital Home-Based Physical Activity Promotion for Older Adults After Total Hip Arthroplasty
Acronym: iPATH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Geriatric Center, Heidelberg University (Unknown); Heidelberg University - Institute of Medical Biometry (IMBI) (Unknown)
Responsible Party: Principal Investigator, Tobias Reiner, Priv.-Doz. Dr. med., University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-324/2024; 1DH2411155 (Other Grant/Funding Number: Dietmar Hopp Foundation)
Record Dates: First submitted 2025-08-07; First posted 2025-08-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Total Hip Arthroplasty (THA); Older Adults (65 Years and Older)
Keywords: Total Hip Arthroplasty; Physical Activity; Older Adults; Digital Intervention; Physical Exercise; Coaching; Patient Education; Postoperative Care; Ambulatory Monitoring; Behavior Change
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, assessor-blinded, three-arm parallel trial with a 12-week intervention period: (1) digital exercise program with personal coaching, (2) digital exercise program without personal coaching, and (3) control group (usual care).
Who Masked: Outcomes Assessor
Masking Description: Biostatistician responsible for data analysis remains blinded until the database is locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Digital exercise program with personal coaching (Intervention Group 1) (Experimental): Participants receive a tablet with the pre-installed training app KOKU, which delivers a 12-week standardized digital home-based strength and balance program. Participants are introduced to KOKU during an initial home visit and are encouraged to complete the program independently over the subsequent 12 weeks. In addition, they receive three individualized coaching sessions via video calls on the tablet during this period. To support self-monitoring and provide feedback on PA behavior - integrated into the BCTs used in the personal coaching - participants also receive a low-cost, easy-to-use wrist-worn activity tracker along with instructions on its use during the initial home visit.
  Interventions: Behavioral: Digital exercise program; Behavioral: Personal coaching for physical activity promotion
- Digital exercise program without personal coaching (Intervention Group 2) (Experimental): Participants receive a tablet with the pre-installed training app KOKU, which delivers a 12-week standardized digital home-based strength and balance program. Participants are introduced to KOKU during an initial home visit and are encouraged to complete the program independently over the subsequent 12 weeks. No personal coaching is provided.
  Interventions: Behavioral: Digital exercise program
- Usual care (Control Group) (No Intervention): Participants receive a tablet without access to the KOKU app and do not receive any personal coaching sessions.

INTERVENTIONS:
Behavioral: Digital exercise program — KOKU is a digital adaptation of the evidence based Otago Exercise Program and Falls Management Exercise program, both designed to improve strength, balance, and reduce fall risk in older adults. KOKU includes 26 balance and strength exercises of varying difficulty. Each exercise is accompanied by written and audio instructions for safe performance and is demonstrated by a virtual trainer. Training sessions consist of three exercises suggested by the KOKU app, which participants are encouraged to perform for as many repetitions as possible until fatigue. Progression is guided by the participant's subjective assessment of effort and difficulty. Participants may choose to perform any exercise at any time, regardless of the app-suggested sequence. The KOKU app also provides reminders to exercise if no activity is detected for two days.
  Arms: Digital exercise program with personal coaching (Intervention Group 1); Digital exercise program without personal coaching (Intervention Group 2)
Behavioral: Personal coaching for physical activity promotion — Personal coaching consists of three video calls conducted via the study tablet by staff trained in BCTs and motivational communication skills. Participants receive a low cost, wrist worn activity tracker during the initial home visit to support self-monitoring and provide feedback on PA behavior. The first virtual coaching session (week 2) focuses on goal setting and action planning, the second session (week 3) addresses identification and management of barriers, and the third session (week 12) serves as a booster to review and adjust activity goals for the post intervention period.
  Arms: Digital exercise program with personal coaching (Intervention Group 1)

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of a 12-week digital home-based intervention program, consisting of a tablet-based exercise program with or without personal coaching, to promote physical activity (PA) in older adults after total hip arthroplasty (THA). The main question it aims to answer is:

• Does the combination of the digital exercise program and personal coaching lead to higher PA six months after THA compared to usual care among older adults?

Secondary questions are:

* Does the digital exercise program alone lead to higher PA compared to usual care?
* Does the digital exercise program combined with personal coaching lead to higher PA compared to the exercise program alone?

Participants' PA will be objectively measured with a body-fixed sensor at 1 week before THA (T1), 6 weeks after THA (T2), and 6 months (i.e. after THA (T3). After the postoperative assessment at T2, participants will be randomly assigned to one of three groups:

* 12-week tablet-based exercise program at home with virtual personal coaching for physical activity promotion
* 12-week tablet-based exercise program at home
* Usual care (control group, no additional intervention)

DETAILED DESCRIPTION:
Hip osteoarthritis is common in older adults and is associated with limitations in activities of daily living, mobility, and quality of life. THA effectively reduces pain and improves physical functioning. However, patients often show no or only minimal increase in their typically low preoperative PA after THA. This lack of PA improvements may result from short rehabilitation periods, persistent sedentary habits, and methodological limitations of PA monitoring methods that focus mainly on frequency or temporal parameters (e.g. step count, walking or active durations).

Digital home-based training programs offer an opportunity for patients to continue structured exercises independently and at flexible times, extending postoperative care beyond standard rehabilitation. In addition, personal coaching that applies behavioral change techniques (BCTs) such as goal setting, action planning, self-monitoring with feedback, and barrier identification and management, may help break sedentary habits and promote PA. Recent advances in wearable sensor technology and processing algorithms now also enable a more detailed monitoring of real-world digital mobility outcomes (DMOs), allowing also capturing spatial-related parameters (e.g., walking distance, stride length, gait speed).

The iPATH study is a three-armed, assessor-blinded, randomized, parallel-group clinical trial evaluating the efficacy of two 12-week digital home-based intervention programs to promote PA in 213 older adults after THA:

1. Digital exercise program with personal coaching (Intervention Group 1)
2. Digital exercise program without personal coaching (Intervention Group 2)
3. Usual care (Control Group) - no additional intervention

Outcome assessments are conducted at 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3; operationally defined as 26 weeks after THA). Randomization occurs after the T2 assessment, which typically coincides with the end of standard inpatient or outpatient rehabilitation. The digital home-based exercise program in the two intervention arms is based on the Keep-On-Keep-Up (KOKU) app, which includes progressive strength and balance exercises to be performed three times per week. Personal coaching includes three virtual sessions designed to promote PA behavior change using BCTs (goal setting, action planning, self-monitoring and feedback [activity tracker], barrier identification and management). Participants in the control group also receive a tablet but have no access to the KOKU app and do not receive any personal coaching sessions.

The primary outcomes are the mean daily step count (first) and mean daily walking distance (second), derived from a body-fixed sensor attached to the participant's lower back for a maximum measurement period of 7 consecutive days using the newest validated processing alogorithms. Secondary outcomes include additional DMOs (e.g., walking duration, number of walking bouts, walking speed, stride length, cadence), life-space mobility, physical capacity, hip pain and function, psychological and cognitive factors (e.g., concerns about falling, executive functioning), falls, intervention adherence and acceptability, health-related resource use, intervention delivery costs, and safety.

The primary study hypothesis is that the combination of the digital exercise program and personal coaching will lead to higher PA six months after THA compared to usual care. Secondary hypotheses are that (1) the digital exercise program alone will increase PA compared to usual care, and (2) the combination of the digital exercise program and personal coaching will increase PA compared to the digital exercise program alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Coxarthrosis with indication for total hip arthroplasty
* Residence within a radius of ≤50 km from Heidelberg
* Ability to walk ≥10 m (with/without walking aid)
* Access to the internet (Wi-Fi) at home
* Written informed consent

Exclusion Criteria:

* Insufficient German language skills
* Insufficient hearing to communicate via (video) telephone
* Insufficient vision to recognize study materials
* Contralateral coxarthrosis with indication for total hip arthroplasty
* Severe medical condition illnesses that compromise physical fitness (heart failure classified as New York Heart Association [NYHA] class ≥3, heart valve defects associated with syncope, cardiac arrhythmia with dizziness, chronic obstructive pulmonary disease [COPD] with oxygen therapy, cancer with chemotherapy and/or radiation, Parkinson's disease with rollator use [Hoehn & Yahr stage ≥4])
* Living in a nursing home
* Planned major medical procedure within the next 6 months with inpatient hospital stay (e.g., further surgery)
* Simultaneous participation in another competing study
* Cognitive impairment (6-item Cognitive Impairment Test [6CIT] score >7 points)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Daily step count | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean daily step count [#/day] is derived from a body-fixed sensor (AX6, Axivity Ltd.) attached to the participant's lower back for a maximum measurement period of 7 consecutive days, using validated processing algorithms.
Daily walking distance | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean daily cumulative walking distance [m/day] is derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms.

SECONDARY OUTCOMES:
Daily walking duration | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean daily walking duration [h/day] derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms.
Daily walking bout count | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean daily walking bout count [#/day] derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms. Mean daily walking bout count is determined for walking bouts >10 s, >30 s, and >60 s.
Daily-life walking bout duration | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean and 90th percentile daily-life walking bout durations [s] derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms.
Daily-life walking speed | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean and 90th percentile daily-life walking speed [m/s] are derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms. Mean and 90th percentile walking speeds are determined for shorter walking bouts (10-30 s) and for longer walking bouts (>30 s).
Daily-life stride length | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean daily-life stride length [cm] is derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms. Mean stride length is determined for shorter (10-30 s) and longer (>30 s) walking bouts.
Daily-life stride duration | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean daily-life stride duration [s] derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms. Mean stride duration is determined for all walking bouts and for longer walking bouts (>30 s).
Daily-life cadence | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Mean and 90th percentile daily-life cadence [steps/min] derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum measurement period of 7 consecutive days, based on validated processing algorithms. Mean cadence is determined for all walking bouts and for longer walking bouts (>30 s), and the 90th percentile cadence for longer walking bouts (>30 s).
Daily-life walking variability | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Bout-to-bout variability [%] in walking bout duration, walking speed and stride length for longer walking bouts (>30 s), cadence and stride duration for all walking bouts, derived from a body-fixed sensor (AX6, Axivity Ltd.) worn on the participant's lower back over a maximum of 7 consecutive days, based on validated processing algorithms.
Physical capacity (a) | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  6-Minute Walk Test (instrumented with the mTEST³ system [mHealth Technologies srl, Bologna, Italy] to capture spatio-temporal gait parameters)
Physical capacity (b) | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Timed Up and Go (instrumented with the mTEST³ system [mHealth Technologies srl, Bologna, Italy] to measure durations of sit-to-walk, walking, turning, and sitting segments)
Physical capacity (c) | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  30-Second Chair Stand Test
Physical capacity (d) | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  4-Meter Gait Speed Test
Hip pain and function | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Oxford Hip Score
Life-space mobility | 1 week preoperatively (T1), and 6 months postoperatively (T3)
  University of Alabama at Birmingham Life-Space Assessment
Concerns about falling | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Short Falls Efficacy Scale-International
Health-related quality of life | 1 week preoperatively (T1) and 6 months postoperatively (T3)
  European Quality of Life 5 Dimensions 5 Level index
Self-perceived health status | 1 week preoperatively (T1) and 6 months postoperatively (T3)
  EuroQol Visual Analogue Scale
Change in self-perceived walking ability | 6 weeks postoperatively (T2) and 6 months postoperatively (T3)
  7-point Global Rating of Change Scale (1= markedly worse, 7 = markedly better)
Self-reported physical activity level | 1 week preoperatively (T1) and 6 months postoperatively (T3)
  University of California Los Angeles Activity Score
Conscientiousness | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Conscientiousness dimension of Big Five Inventory-2
Exercise motivation | 1 week preoperatively (T1), 6 weeks postoperatively (T2), and 6 months postoperatively (T3)
  Behavioural Regulation in Exercise Questionnaire
Rate of falls | From 6 weeks postoperatively (T2) to 6 months postoperatively (T3)
  Daily fall calendars
Executive functioning | 1 week preoperatively (T1) and 6 months postoperatively (T3)
  Trail Making Test A & B
Health-related resource use | 1 week preoperatively (T1) and 6 months postoperatively (T3)
  Questionnaire for Health-Related Resource Use in an Elderly Population

OTHER OUTCOMES:
Adverse events | 6 weeks postoperatively (T2) and 6 months postoperatively (T3); interim events recorded as reported.
  Frequency, type, severity, and relation to the intervention of participant-reported (serious) adverse adverse events will be documented using standardized case report forms.
Training adherence (a) | 6 months postoperatively (T3)
  Exercise Adherence Rating Scale
Training adherence (b) | 6 months postoperatively (T3)
  Usage data of the training app (KOKU) retrieved from the tablet
Intervention acceptability (a) | 6 months postoperatively (T3)
  Theoretical Framework of Acceptability Questionnaire (range: 7-35 points, higher scores indicate higher acceptability)
Intervention acceptability (b) | 6 months postoperatively (T3)
  5-point Likert scale on global acceptability (1 = completely unacceptable, unacceptable, 5 = completely acceptable)
Intervention delivery costs | From the start of the intervention to the end of the intervention (up to 12 weeks)
  Intervention costs [€] derived from personnel, material, and travel expenses, using standardized national unit costs.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Reiner, PhD, MD, Principal Investigator — Department of Orthopaedics, Heidelberg University Hospital; Christian Werner, PhD, Principal Investigator — Geriatric Center, Heidelberg University
Locations (1):
- Department of Orthopaedics, Heidelberg University Hospital, Heidelberg, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
In line with the principles of open science, anonymized individual participant data from the iPATH trial will be made available to qualified researchers after the primary evaluation has been completed and published. Data will be shared in a format that does not permit identification of individual participants and in full compliance with applicable data protection regulations (e.g., General Data Protection Regulation, EU data protection standards). Access to the data will be provided via a recognized open-access repository and require a formal application with a description of the proposed research project.
Supporting Information: Study Protocol, SAP
Time Frame: Anonymized individual participant data (IPD) will be made available approximately 6 months after publication of the primary evaluation results and will remain accessible without a predefined end date.
  The study protocol will be submitted for publication in an open-access, peer-reviewed journal before the last patient is enrolled.
  The statistical analysis plan (SAP) will be published alongside the primary evaluation results.
Access Criteria: Access will be granted to qualified researchers affiliated with recognized academic or research institutions. A formal application including a research proposal is required, and applicants must agree to a data use agreement ensuring ethical use and compliance with EU data protection regulations. Approved applicants will access the data via the designated open-access repository.